CLINICAL TRIAL: NCT00420511
Title: A Randomized Controlled Pilot Study Assessing the Effect of Sitagliptin on the Preservation of Beta-Cell Function in Patients With Type 2 Diabetes
Brief Title: Beta-Cell Function and Sitagliptin Trial (BEST)
Acronym: BEST
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Bernard Zinman, Director, Leadership Sinai Centre for Diabetes, Samuel Lunenfeld Research Institute, Mount Sinai Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 065-00
Record Dates: First submitted 2007-01-10; First posted 2007-01-11 (Estimated); Results first posted 2011-12-29 (Estimated); Last update posted 2012-01-02 (Estimated); Status verified 2011-12

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 diabetes; beta-cell function; sitagliptin; intensive insulin therapy
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate; Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sitagliptin (Experimental): Sitagliptin 100mg once a day (od) by mouth (po)
  Interventions: Drug: Sitagliptin; Drug: metformin
- Placebo arm (Placebo Comparator): Placebo once a day (od) by mouth (po)
  Interventions: Drug: Placebo; Drug: metformin

INTERVENTIONS:
Drug: Sitagliptin — sitagliptin 100 mg once a day
  Other Names: januvia
  Arms: Sitagliptin
Drug: Placebo — placebo once a day
  Arms: Placebo arm
Drug: metformin — metformin 1000 mg twice a day (bid) by mouth (po)
  Other Names: glucophage

SUMMARY:
Type 2 diabetes mellitus (T2DM) is a chronic metabolic disorder characterized by progressive deterioration in the function of the pancreatic beta-cells, which are the cells that produce and secrete insulin (the hormone primarily responsible for the handling of glucose in the body). The investigators propose a double-blind, randomized controlled pilot study comparing the effect of sitagliptin (a novel anti-diabetic drug with beta-cell protective potential) versus placebo, on the preservation of beta-cell function over one year in patients with T2DM on metformin, the first-line agent for the treatment of T2DM (ie. the study groups will be (i) sitagliptin and metformin versus (ii) placebo and metformin). This study may demonstrate an important beta-cell protective capacity of sitagliptin.

Hypothesis: In patients with T2DM on metformin, treatment with the DPP-IV inhibitor sitagliptin will preserve pancreatic beta-cell function.

DETAILED DESCRIPTION:
Medications currently used in the treatment of T2DM have not been shown to modify the progressive decline in beta-cell function that occurs over time. Recent evidence, however, suggests that a new class of anti-diabetic medications, called dipeptidyl peptidase-IV (DPP-IV) inhibitors, may be able to protect beta cells and hence alter the natural history of T2DM. We thus wish to study the effect of sitagliptin (a DPP-IV inhibitor) on the preservation of beta-cell function in patients with T2DM randomized to either (i) sitagliptin and metformin or (ii) placebo and metformin.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women between the ages of 30 and 75 inclusive
2. Physician-diagnosed type 2 diabetes on 0-2 oral hypoglycemic agents
3. Negative for anti-glutamic acid decarboxylase (anti-GAD_ antibodies (to rule out Latent Autoimmune Diabetes of Adults (LADA)
4. A1c at screening between 6.5% and 9% inclusive if on no oral hypoglycemic agents or 6.0% and 9.0% inclusive if on 1-2 oral hypoglycemic agents

Exclusion Criteria:

1. Current insulin therapy
2. Type 1 diabetes or secondary forms of diabetes
3. Any major illness with a life expectancy of < 5 years or that may interfere with the patient's participation in the study
4. Involvement in any other study requiring drug therapy
5. Renal dysfunction as evidenced by serum creatinine >/= 136 umol/L for males or >/= 124 umol/L for females or abnormal creatinine clearance (< 60 ml/min by Modification of Diet in Renal Disease (MDRD) formula)
6. Hepatic disease considered to be clinically significant (includes jaundice, chronic hepatitis, or previous liver transplant) or transaminases > 2.5 times the upper limit of normal
7. Excessive alcohol consumption, defined as > 14 alcoholic drinks per week for males and > 9 alcoholic drinks per week for females
8. Pregnancy or unwillingness to use reliable contraception. Women should not be planning pregnancy for the duration of the study. Reliable contraception includes: birth control pill, intra-uterine device, abstinence, tubal ligation, partner vasectomy, or condoms with spermicide. Any women who miss a menstrual period or think that they may be pregnant must have a pregnancy test as soon as possible
9. History of serious arrhythmia or atrioventricular block on baseline electrocardiogram
10. Uncontrolled hypertension (systolic blood pressure > 180 mm Hg or diastolic blood pressure > 110 mm Hg)
11. Unwillingness to undergo multiple daily insulin injection therapy for 4 weeks
12. Unwillingness to perform capillary blood glucose monitoring at least 4 times per day during intensive insulin therapy

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2007-01; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Zinman, MD, Principal Investigator — Leadership Sinai Centre for Diabetes, University of Toronto; Ravi Retnakaran, MD, Principal Investigator — Leadership Sinai Centre for Diabetes, University of Toronto
Locations (1):
- Leadership Sinai Centre for Diabetes, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Stein CM, Kramer CK, Zinman B, Choi H, Opsteen C, Retnakaran R. Clinical predictors and time course of the improvement in beta-cell function with short-term intensive insulin therapy in patients with Type 2 diabetes. Diabet Med. 2015 May;32(5):645-52. doi: 10.1111/dme.12671. Epub 2015 Jan 7. PMID 25495067

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from outpatient clinics at the Leadership Sinai Centre for Diabetes between February 2007 and October 2008.
Pre-assignment Details: Participants underwent prerandomization phase of 4-8 weeks of intensive insulin therapy (IIT) consisting of basal detemir and premeal insulin aspart. Only participants who achieved fasting glucose <7.0 mmol/L 1 day after completing IIT were randomized to either sitagliptin 100 mg once daily or matching placebo.
Groups:
- Sitagliptin: Sitagliptin 100 mg once daily and metformin 1000 mg twice a day (bid) by mouth po
- Placebo: Matching placebo once daily and metformin 1000 mg twice a day (bid) by mouth (po)
Period: Overall Study
Arm/Group | Sitagliptin | Placebo
Started | 10 | 11
Completed | 8 | 10
Not Completed | 2 | 1
Not completed — Adverse Event | 1 | 1
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sitagliptin | Placebo | Total
Number analyzed (Participants) | 10 | 11 | 21
Age Continuous [Median (Inter-Quartile Range); unit: years] | 61.3 [45.5 to 69.5] | 60.8 [51.3 to 61.4] | 60.9 [47.9 to 61.4]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 6 | 8 | 14
Race/Ethnicity, Customized [Number; unit: participants]
  White | 4 | 9 | 13
  Other | 6 | 2 | 8
Body Mass Index [Median (Inter-Quartile Range); unit: kg/m^2] | 34.3 [27.3 to 42.6] | 32.7 [31.0 to 41.1] | 32.7 [28.6 to 41.5]
Duration of diabetes [Median (Inter-Quartile Range); unit: years] | 2.8 [2.0 to 4.0] | 3.5 [2.0 to 8.0] | 3.0 [2.0 to 6.0]
HbA1c [Median (Inter-Quartile Range); unit: percent glycosylated hemoglobin] | 6.2 [5.8 to 6.9] | 6.1 [5.9 to 6.9] | 6.1 [5.8 to 6.9]
Area-Under-The-Curve (C-peptide/glucose) / HOMA-IR [Median (Inter-Quartile Range); unit: index of beta-cell function] — Area-under-the-C-peptide-curve (AUCCpep) and area-under-the-glucose-curve (AUCgluc) from 0 to 240 minutes during meal tests were calculated by trapezoidal rule. Insulin resistance was assessed by Homeostasis Model Assessment of Insulin Resistance (HOMA-IR). Beta-cell function was assessed using the ratio of AUCCpep to AUCgluc divided by HOMA-IR (AUCCpep/gluc/HOMA-IR), a measure of insulin secretion in the context of ambient insulin sensitivity, analogous to the disposition index and Insulin Secretion-Sensitivity Index-2 (ISSI-2). Higher AUCCpep/gluc/HOMA-IR indicates better beta-cell function.
  index of beta-cell function | 114.8 [76.3 to 208.7] | 126.0 [79.8 to 159.8] | 120.0 [66.3 to 129.6]

OUTCOME MEASURES:

1. Primary Outcome: Preservation of Beta-cell Function Measured by Area-under-the-curve (C-peptide/Glucose)/HOMA-IR
Description: Area-under-the-C-peptide-curve (AUCCpep) and area-under-the-glucose-curve (AUCgluc) from 0 to 240 minutes during meal tests were calculated using the trapezoidal rule. Insulin resistance was assessed using the Homeostasis Model Assessment of Insulin Resistance (HOMA-IR). Beta-cell function was assessed using the ratio of total AUCCpep to AUCgluc divided by HOMA-IR (AUCCpep/gluc/HOMA-IR), a measure of insulin secretion in the context of ambient insulin sensitivity, analogous to the disposition index and adaptation index. Higher AUCCpep/gluc/HOMA-IR is indicative of better beta-cell function.
Time Frame: 48 weeks
Measure: Median (Inter-Quartile Range); unit: index of beta-cell function
Groups:
- Sitagliptin: Sitagliptin 100 mg once daily and metformin 1000 mg twice a day (orally administered)
- Placebo: Matching placebo once daily and metformin 1000 mg twice a day (orally administered)
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 10 | 11
index of beta-cell function | 80.4 [52.5 to 205.6] | 71.2 [40.3 to 139.8]

2. Secondary Outcome: Insulinogenic Index Divided by HOMA-IR at 48 Weeks
Description: Insulinogenic index was calculated as the incremental change in insulin from 0 to 30 minutes divided by the incremental change in glucose over the same period of time. Insulinogenic index divided by HOMA-IR provides an additional measure of beta-cell function. A higher value indicates better beta-cell function
Time Frame: 48 weeks
Measure: Median (Inter-Quartile Range); unit: index of beta-cell function
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 10 | 11
index of beta-cell function | 3.9 [1.9 to 4.9] | 1.8 [1.3 to 2.8]

3. Secondary Outcome: Fasting Blood Glucose at 48 Weeks
Time Frame: 48 weeks
Measure: Median (Inter-Quartile Range); unit: mmol/l
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 10 | 11
mmol/l | 6.9 [5.5 to 7.4] | 6.7 [6.0 to 7.9]

4. Secondary Outcome: Area-under-the-glucose-curve (AUCglucose) on Meal Test at 1 Year
Time Frame: 1 year
Reporting Status: Not Posted

5. Secondary Outcome: Time to Loss of Glycemic Control
Time Frame: 1 year
Reporting Status: Not Posted

6. Secondary Outcome: Proportion of Patients Achieving Sustained Normoglycemia Off Medication at 1-week Post-insulin Therapy
Time Frame: 1 year
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Sitagliptin | Placebo
Serious Adverse Events (participants affected / at risk) | 1/10 | 1/11
Other Adverse Events (participants affected / at risk) | 0/10 | 0/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sitagliptin (N=10) | Placebo (N=11)
Generalized rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Renal tumor (Renal and urinary disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The modest sample size of this pilot study may have lacked sufficient statistical power to detect an effect on preservation of beta-cell function.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No